CLINICAL TRIAL: NCT04852471
Title: Improving Quality of Life Using Patient Reported Outcomes Measures Post-operative Via Text Messaging: a Randomized Control Trial (PROMPT Study)
Brief Title: Improving Quality of Life Using Patient Reported Outcomes Measures Post-operative Via Text Messaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2020.173; HUM00190175 (Other: University of Michigan)
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Gynecologic Cancer
Keywords: laparotomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Post-Operative Counseling + FACT-G (Control Arm) (Active Comparator): Patients will receive the standard postoperative counseling at discharge, discharge instructions, and the link to website with postoperative instructions. Patients will complete the Functional Assessment of Cancer Therapy - General (FACT-G).
  Interventions: Behavioral: Standard Post-Operative Counseling + FACT-G
- Standard Post-Operative Counseling + PROM survey + FACT-G (Intervention Arm) (Experimental): Patients will receive the standard postoperative counseling at discharge, discharge instructions, and the link to website with postoperative instructions. The intervention arm will receive and complete the Patient-Reported Outcome Measure (PROM) survey via the SMS text messaging service on a set schedule. Patients will complete the FACT-G.
  Interventions: Behavioral: Standard Post-Operative Counseling + FACT-G; Behavioral: PROM symptom tracker

INTERVENTIONS:
Behavioral: Standard Post-Operative Counseling + FACT-G — Counseling at discharge + FACT-G at enrollment, at 15-18 and at 30-32 days post-operative.
Behavioral: PROM symptom tracker — A 12-item symptom tracker adopted from the Patient Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (NCI-PRO-CTCAE), delivered via text, on days 4, 6, 8, 12, 18, 24, and 30 post surgery.
  Arms: Standard Post-Operative Counseling + PROM survey + FACT-G (Intervention Arm)

SUMMARY:
This study is investigating a new way to monitor patients who are recovering at home after surgery. This study uses text messages to ask patients to review their own symptoms and then reply with the level of severity of specific symptoms. Based on each patient's specific response to the text message survey, a pre-programmed, automated response will be sent from the study prompting the patient to take specific actions (or no action if no symptoms). Investigators will assess whether this method improves patients' well-being as compared to the current standard of care for patients. Currently, after surgery, patients are provided counseling and written instructions when they leave the hospital on how to care for themselves at home. If the patient has questions or concerns, they contact their care team. The optimal way to help patients assess their own symptoms at home remains unknown. Investigators are also assessing if using the symptom survey reduces readmissions to the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or greater.
* Planning to undergo a surgical procedure via a laparotomy incision for a suspected or known gynecologic malignancy. There is no restriction on the spectrum of pathology or disease.
* The ability and willingness to send and receive short messaging service (SMS) text messages.
* Able to read and understand English.
* Willing and able to provide informed consent

Exclusion Criteria:

* Persons who are planning to undergo a minimally invasive procedure without laparotomy.
* Persons unable to be contacted by SMS text message or choose to opt-out of the study.
* Patients who do not have access to the internet via a home computer or a smart phone.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Mean total score on FACT-G | 30-32 days post-operative
  The mean total score on the FACT-G will be compared between the two arms. The FACT-G is a 27-item questionnaire that covers four HR-QOL sub-domains: physical, social, emotional, and functional well-being. Each of the questions will be scored on a scale from 0 (Not at all) to 4 (Very much) using a manual scoring template in which some items are reverse scored. The minimally important difference (MID) is 5 points for the FACT-G questionnaire. In other words, five points is the most minimal difference between the control group and treatment group scores that would indicate a clinically meaningful change. A positive change in points indicates better QOL.

SECONDARY OUTCOMES:
Proportion of patients who had non-standard clinic visits | 30 days post-operative
  The proportion of patients who are seen in the clinic for visits other than a scheduled post-operative visit. Data collected by chart review.
Proportion of patients who called the care team | 30 days post-operative
  Data collected by chart review.
Proportion of patients seen in urgent care clinics | 30 days post-operative
  Data collected by chart review.
Proportion of patients seen in emergency room | 30 days post-operative
  Data collected by chart review.
Proportion of patients readmitted to hospital | 30 days post-operative
  Data collected by chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Shitanshu Uppal, MBBS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No